CLINICAL TRIAL: NCT06311825
Title: The Effect of Horticultural Therapy on Loneliness and Life Satisfaction in Elderly Adults Living in Nursing Home
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Dilara Haktanır, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstanbulUCDH
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Horticultural Therapy; Loneliness; Satisfaction, Personal; Aging
Keywords: Horticultural Therapy; Elderly; Loneliness; Life Satisfaction
MeSH Terms: conditions — Personal Satisfaction | interventions — Horticultural Therapy

STUDY DESIGN:
Intervention Model Description: Two parallel groups randomized control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horticultural Therapy Group (Experimental) (Experimental): Horticultural therapy will be applied to experimental group.
  Interventions: Other: Horticultural Therapy
- Controls (Control Group) (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Horticultural Therapy — One week before horticultural therapy (HT) interventions, face-to-face interviews will be held with the individuals in the experimental group and the forms will be filled in as a pretest.
  HT will be applied to the experimental group. The application period was determined as a total of 6 weeks with 50-minute sessions twice a week.
  Before starting the HT sessions, area preparations will be made and a safe therapeutic garden will be established.
  Medicinal and aromatic plants will be selected that can grow in Turkey, are not harmful to human health, are fragrant and colorful in order to stimulate the senses, and according to air temperature and physical conditions.
  HT sessions will consist of gardening activities (group meeting, introduction of plants and cultivation).
  After HT interventions, the forms will be filled as a post test. The forms will be filled again 4 weeks after the end of the interventions for follow-up.
  Arms: Horticultural Therapy Group (Experimental)

SUMMARY:
Loneliness in elderly individuals increases with age and negatively affects individuals by decreasing life satisfaction. In recent years, horticultural therapy is a type of therapy that has developed and is added routine care of elderly individuals living in nursing homes. Social interaction, life satisfaction, feelings of success and responsibility and increase while loneliness and depression levels decrease through human-nature interaction in horticultural therapy.

In our country, no study has been found on the effects of horticultural therapy on physical or mental health in elderly individuals. This research will be conducted as a randomized control group study to examine the effects of horticultural therapy on loneliness and life satisfaction in elderly individuals living in nursing homes.

DETAILED DESCRIPTION:
In recent years, the elderly population is increasing in Turkey and around the world. In our country from 2002 to 2022, the number of elderly people receiving care increased 2.8 times. Elderly individuals frequently complain about loneliness and think that they are abandoned. Loneliness is a multidimensional concept consisting of emotional loneliness and social loneliness, and reported that it reduces life satisfaction in elderly individuals.

There are many non pharmacological applications aimed at reducing loneliness and increasing life satisfaction however in recent years, the use of horticultural therapy in the world has attracted attention. In horticultural therapy interventions, gardening activities are carried out using indoor and outdoor plants. The plants which is medicinal and aromatic selected according to culture and cultivation. The plants contribute to the improvement of physical and mental health by stimulating 5 senses that visual, hearing, tasting, touching and smell.

Horticultural therapy is important in terms of providing social activity, reducing loneliness and increasing life satisfaction in elderly individuals using the healing power of nature.

Horticultural therapy is also used by nurses who are mental health professionals. In Turkey, there is no study to examine effects of horticultural therapy effects on mental health in elderly individuals. It is thought that with this study, it will be important to apply a new method in our country and contribute to nursing science in non-pharmacological applications.

ELIGIBILITY:
Inclusion Criteria:

* Over 60 years old,
* Being literate,
* Living in nursing home for at least 3 months,
* Not diagnosed with dementia,
* Mini Mental Test Score>24
* No additional neurological disease,
* No history of serious psychiatric illness,
* Not in the acute phase of a systemic disease,
* No vision or hearing loss that would hinder gardening activities,
* Does not have a physical disability that would hinder gardening activities,
* No history of falls,
* Not participating in different applications at the same time.

Exclusion Criteria:

* Does not meet the inclusion criteria,
* Persons with allergic reactions to soil and plants that may hinder with gardening activities.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Loneliness Scale for Elderly | 3 Month
  The scale measures the loneliness levels of the elderly and consists of 11 items. The scale consists of two sub-dimensions: social loneliness and emotional loneliness. In the scale, 5 items are coded directly (1, 4, 7, 8, 11), and 6 items are reverse coded (2, 3, 5, 6, 9, 10). The degree to which the person experiences the situation contained in each statement in the scale is determined by a 3-point Likert type rating (0 = yes, 1 = possible, 2 = no). The lowest score to be obtained from the scale is 0 and the highest score is 22. Higher scale scores indicate increased loneliness levels. The internal consistency Cronbach's alpha coefficient is α=is .85.
Life Satisfaction Scale | 3 Month
  The scale consists of 5 items and a single sub-dimension. The original scale is a seven-point Likert type, with answers ranging from 1-Strongly Agree to 7-Strongly Disagree. In the Turkish validity and reliability study conducted on adults, the seven-point Likert type was not found to be suitable for Turkish culture and the number of steps was reduced from seven to five. Scoring of the items in the scale; It was determined as "I totally disagree (1), I slightly agree (2), I moderately agree (3), I largely agree (4) and I totally agree (5)". The Cronbach Alpha internal consistency coefficient of the scale was reported as 0.88 and the test-retest reliability was reported as 0.97.

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Bilgin, PhD, Study Director — Istanbul University - Cerrahpasa; Sima Pouya, PhD, Study Director — Malatya Inonu University
Locations (1):
- Istanbul University - Cerrahpasa (IUC), Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No